CLINICAL TRIAL: NCT03676348
Title: Health Related Quality of Life in Thyroid Cancer Patients, and in Patients With Thyroid Nodules Suspicious of Cancer
Brief Title: HRQOL in Thyroid Cancer and Thyroid Tumours
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Bianca M.R. Lorntzsen, MD, PhD candidate, Oslo University Hospital
Other Study IDs: 2017/1040
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Thyroid Nodule; Thyroid Cancer; Quality of Life
Keywords: quality of life; health related quality of life; thyroid cancer; thyroid nodule; thyroid neoplasm; thyroid surgery; patient reported outcome measurements
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Most patients with thyroid cancer have a long life expectancy, and it has been assumed among health professionals that therefore the quality of life (QOL) is good. Some European studies have shown that the quality of life among thyroid cancers is worse than the general population, and almost as low as other cancer diagnoses, with a worse prognosis and a more burdening treatment.

Aim: To examine prospectively the quality of life in participants undergoing diagnostic thyroid surgery and participants undergoing surgery for certain thyroid cancer. By examining both groups we wish to find answers if quality of life is affected, and if so - mostly affected by the diagnosis or the surgery itself.

Methods: Participants enroll the study after informed consent, and quality of life will be assessed using quality of life questionnaires EORTC QLQ C30, EORTC THY 47 and EORTC FA12 before surgery, and 6 and 12 months after surgery. This study will form two main groups of participants; with and without thyroid cancer.

DETAILED DESCRIPTION:
Most patients with thyroid cancer have a long life expectancy, and it has been assumed among health professionals that therefore the quality of life (QOL) is good. Some European studies have shown that the QOL among thyroid cancers is worse than the general population, and almost as low as other cancer diagnoses, with a worse prognosis and a more burdening treatment.

This study aims to examine the quality of life in patients undergoing diagnostic surgery for thyroid tumour(s), or thyroid surgery as part of a cancer treatment.

Participants will undergo standard work up and treatment for their thyroid tumour(s). Clinical data will be extracted from medical records at Oslo University Hospital (OUH). Questionnaires on Health related quality of life (HRQOL) are be filled out before surgery and at follow up visits at 6 and 12 months after surgery. Participants that do not meet at follow-up, will receive the questionnaires by mail.

At the end of the study there will be three subgroups of participants: (a) Benign tumour, (b) Malignant tumour with radioiodine treatment, (c) Malignant tumour without radioiodine treatment.

Questionnaires from European Organization for Research and Treatment of Cancer (EORTC) will be used, as they are well validated and relatively widely used. The EORTC QLQ C30 was chosen for a general view on HRQOL, as well as an available Norwegian general population for comparison. For a more disease specific questionnaire, the EORTC THY47 is used, a module of EORTC QLQ C30 on thyroid cancer. In addition we wish to capture a possibly important element in participants undergoing thyroid surgery, and where a fraction of participants may be hypothyroid for a period of time - therfore a fatigue module, the EORTC FA12 was added.

Calculations on sample size were performed by statistician R Sørum Falk at the Centre of Biostatistics and Epidemiology of Oslo University Hospital.

Intraobserver analysis of plotting and calculations is planned.

ELIGIBILITY:
Inclusion Criteria:

* planned hemi- or total thyroidectomy at the ENT-Department of Oslo University Hospital
* tumour in the thyroid gland With fine needle aspiration results of Bethesda 3-6, or other clinical manifestations suspicious of cancer.
* ability to understand and Complete the quesitionnaires
* informed consent to participation

Exclusion Criteria:

* unable to Complete or understand the questionnaires
* age below 18 years
* thyroid surgery within the last 2 years
* thyroid surgery on other indications than listed above
* participants With postoperative external radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oslo University Hospital (OUH) is a regional hospital. The Ear Nose and Throat (ENT) department is sharing the responsibility for diagnosis and treatment of thyroid cancer with one other location within OUH. Patients planned for thyroid surgery at the ENT department of OUH , will be asked to participate in the study. At the point of recruitment to the study, the final diagnosis in unknown for the doctor as well as the participant, as the result will come from histopathologcal examination of the surgery specimen. Participants will undergo standard work up for their thyroid tumour(s), and standard treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change in global HRQOL score | Circa 12 months from date of (last) thyroid surgery for the individual participant
  Change in global HRQOL score between start and at 12 months postoperatively after thyroid surgery. A change of more than 10% is set as a limit for a significant change.

SECONDARY OUTCOMES:
Change in fatigue score | Circa 12 months from date of (last) thyroid surgery for the individual participant
  Change in fatigue score between start and at 12 months postoperatively after thyroid surgery. A change of more than 10% is set as a limit for a significant change.
Change in HRQOL before and after radioiodine treatment | Circa 12 months from date of (last) thyroid surgery for the individual participant
  Change in HRQOL before and after radioiodine treatment.
Change in HRQOL between participants With benign and malignant tumours | Circa 12 months from date of (last) thyroid surgery for the individual participant
  Change in HRQOL between participants With benign and malignant tumours.

CONTACTS AND LOCATIONS:
Overall Officials: Terje A Osnes, MD, PhD, Principal Investigator — Professor otorhinolaryngology, Rikshospitalet, Oslo University Hospital. Head of department, otorhinolaryngology - head and neck surgery, Rikshospitalet, Oslo University Hospital
Locations (1):
- ENT department, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No